CLINICAL TRIAL: NCT05019430
Title: Behavioral Effects of Drugs (Inpatient): 42 (Cocaine and Zolmitriptan)
Brief Title: Cocaine and Zolmitriptan
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: William Stoops (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, William Stoops, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BED In 42; R01DA052203 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-24 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Cocaine; zolmitriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo. Cocaine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Cocaine; Drug: Placebo oral capsule
- Zolmitriptan Dose 1 (Experimental): Subjects will be maintained on oral zolmitriptan dose 1. Cocaine will be administered acutely during zolmitriptan dose 1 maintenance. Placebo will be administered acutely during zolmitriptan dose 1 maintenance.
  Interventions: Drug: Cocaine
- Zolmitriptan Dose 2 (Experimental): Subjects will be maintained on oral zolmitriptan dose 2. Cocaine will be administered acutely during zolmitriptan dose 2 maintenance. Placebo will be administered acutely during zolmitriptan dose 2 maintenance.
  Interventions: Drug: Cocaine; Drug: Zolmitriptan
- Zolmitriptan Dose 3 (Experimental): Subjects will be maintained on oral zolmitriptan dose 3. Cocaine will be administered acutely during zolmitriptan dose 3 maintenance. Placebo will be administered acutely during zolmitriptan dose 3 maintenance.
  Interventions: Drug: Cocaine; Drug: Zolmitriptan

INTERVENTIONS:
Drug: Cocaine — The pharmacodynamic effects of cocaine will be determined during maintenance on placebo and zolmitriptan.
Drug: Placebo oral capsule — The pharmacodynamic effects of placebo will be determined.
  Arms: Placebo
Drug: Zolmitriptan — The pharmacodynamic effects of zolmitriptan maintenance will be determined.
  Arms: Zolmitriptan Dose 2; Zolmitriptan Dose 3

SUMMARY:
Cocaine potently inhibits the reuptake of serotonin (5-HT). Increased synaptic 5-HT resulting from this reuptake inhibition activates multiple 5-HT receptor subtypes. Some of these receptor subtypes have been implicated in the abuse-related effects of cocaine, including its primary reinforcing effects (i.e., cocaine taking behavior). 5-HT1b receptors, which are autoreceptors on 5-HT nerve endings that regulate 5-HT release and heteroreceptors that also mediate other neurotransmitter release, play a particularly important role in cocaine effects, likely because they are highly expressed in the mesocorticolimbic system. The 5-HT1b system displays profound dysregulation during both active cocaine use and abstinence. Initial preclinical research showed that selective 5-HT1b agonists enhanced the reinforcing and locomotor effects of cocaine during ongoing cocaine administration, but subsequent research showed that these agents robustly attenuated reinstatement of cocaine- and cue-primed cocaine seeking behavior. These findings have been replicated in rigorously conducted studies using multiple schedules of reinforcement and negative sucrose reinforcement controls across laboratories. Notably, though, these preclinical studies used compounds not approved for use in humans, hindering translation. Recently published data show that zolmitriptan, a commercially available selective 5-HT1b agonist migraine medication, also selectively attenuates the reinforcing and other abuse-related effects of cocaine, regardless of stage of use (i.e., ongoing or extinguished cocaine self-administration).

Although a robust preclinical literature supports the premise that 5-HT1b activation reduces a number of cocaine-associated behaviors (e.g., self-administration, cocaine seeking), this area remains unstudied in humans. The overarching goal of this project is to advance these promising preclinical findings, specifically those with zolmitriptan, to a clinical population, thereby demonstrating that the 5-HT1b system plays a key role in the effects of cocaine in humans

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance use disorder that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine or zolmitriptan

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: This study used a within subjects design (i.e., all subjects were to receive all oral zolmitriptan maintenance conditions [0, 2.5, 5 and 10 mg] and intravenous cocaine doses [0, 10 and 30 mg/70 kg]). Nine subjects completed the full study. Three additional subjects were enrolled but discharged prior to completing the full study. Data from completed sessions for those subjects are included here.
  Dose Condition 1: 0 mg zolmitriptan, 0 mg cocaine Dose Condition 2: 0 mg zolmitriptan, 10 mg cocaine Dose Condition 3: 0 mg zolmitriptan, 30 mg cocaine Dose Condition 4: 2.5 mg zolmitriptan, 0 mg cocaine Dose Condition 5: 2.5 mg zolmitriptan, 10 mg cocaine Dose Condition 6: 2.5 mg zolmitriptan, 30 mg cocaine Dose Condition 7: 5 mg zolmitriptan, 0 mg cocaine Dose Condition 8: 5 mg zolmitriptan, 10 mg cocaine Dose Condition 9: 5 mg zolmitriptan, 30 mg cocaine Dose Condition 10: 10 mg zolmitriptan, 0 mg cocaine Dose Condition 11: 10 mg zolmitriptan, 10 mg cocaine Dose Condition 12: 10 mg zolmitriptan, 30 mg cocaine
Period: Overall Study
Arm/Group | Overall Study
Started | 12
Dose Condition 1 | 9
Dose Condition 2 | 10
Dose Condition 3 | 10
Dose Condition 4 | 10
Dose Condition 5 | 10
Dose Condition 6 | 10
Dose Condition 7 | 11
Dose Condition 8 | 11
Dose Condition 9 | 11
Dose Condition 10 | 11
Dose Condition 11 | 11
Dose Condition 12 | 11
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: This study used a within subjects design (i.e., all subjects were to receive all oral zolmitriptan maintenance conditions [0, 2.5, 5 and 10 mg] and intravenous cocaine doses [0, 10 and 30 mg/70 kg]). Ten subjects completed the full study. Two additional subjects were enrolled but discharged prior to completing the full study. Data from completed sessions for those subjects are included here.
Arm/Group | Overall Study
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Reinforcing Effects of Cocaine
Description: Number of Times Subjects Choose Cocaine (Maximum of 5 Choices) Over Money
Time Frame: Over approximately four hours on each experimental session day, which generally occurred on Days 5-7, 13-15, 21-23 and 29-31 of inpatient admission.
Population: Subjects completing the dose condition
Measure: Mean (Standard Deviation); unit: number of times subjects chose cocaine
Groups:
- Dose Condition 1: 0 mg/70 kg IV Cocaine and 0 mg/day Oral Zolmitriptan
- Dose Condition 2: 10 mg/70 kg IV Cocaine and 0 mg/day Oral Zolmitriptan
- Dose Condition 3: 30 mg/70 kg IV Cocaine and 0 mg/day Oral Zolmitriptan
- Dose Condition 4: 0 mg/70 kg IV Cocaine and 2.5 mg/day Oral Zolmitriptan
- Dose Condition 5: 10 mg/70 kg IV Cocaine and 2.5 mg/day Oral Zolmitriptan
- Dose Condition 6: 30 mg/70 kg IV Cocaine and 2.5 mg/day Oral Zolmitriptan
- Dose Condition 7: 0 mg/70 kg IV Cocaine and 5 mg/day Oral Zolmitriptan
- Dose Condition 8: 10 mg/70 kg IV Cocaine and 5 mg/day Oral Zolmitriptan
- Dose Condition 9: 30 mg/70 kg IV Cocaine and 5 mg/day Oral Zolmitriptan
- Dose Condition 10: 0 mg/70 kg IV Cocaine and 10 mg/day Oral Zolmitriptan
- Dose Condition 11: 10 mg/70 kg IV Cocaine and 10 mg/day Oral Zolmitriptan
- Dose Condition 12: 30 mg/70 kg IV Cocaine and 10 mg/day Oral Zolmitriptan
Arm/Group | Dose Condition 1 | Dose Condition 2 | Dose Condition 3 | Dose Condition 4 | Dose Condition 5 | Dose Condition 6 | Dose Condition 7 | Dose Condition 8 | Dose Condition 9 | Dose Condition 10 | Dose Condition 11 | Dose Condition 12
Number analyzed (Participants) | 9 | 10 | 10 | 10 | 10 | 10 | 11 | 11 | 11 | 11 | 11 | 11
number of times subjects chose cocaine | 1.4 (1.96) | 4 (1.61) | 4.5 (1.51) | 0.7 (1.57) | 3.6 (2.06) | 4.5 (1.58) | 0.6 (1.57) | 3.5 (1.97) | 4.6 (0.67) | 0.7 (1.42) | 4.1 (1.45) | 4.2 (1.83)

ADVERSE EVENTS:
Time Frame: Approximately 1 month of inpatient admission.
Description: Definitions for adverse events/serious adverse events follow clinicaltrials.gov guidelines.
Groups:
- Zolmitriptan (0 mg/Day): Maintenance on 0 mg Zolmitriptan/day
- Zolmitriptan (2.5 mg/Day): Maintenance on 2.5 mg Zolmitriptan/day
- Zolmitriptan (5 mg/Day); Zolmitriptan (10 mg/Day): Maintenance on 5 mg Zolmitriptan/day
Arm/Group | Zolmitriptan (0 mg/Day) | Zolmitriptan (2.5 mg/Day) | Zolmitriptan (5 mg/Day) | Zolmitriptan (10 mg/Day)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 11/11 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolmitriptan (0 mg/Day) (N=10) | Zolmitriptan (2.5 mg/Day) (N=10) | Zolmitriptan (5 mg/Day) (N=11) | Zolmitriptan (10 mg/Day) (N=11)
Blood clot (Blood and lymphatic system disorders) | 1 (1) | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolmitriptan (0 mg/Day) (N=10) | Zolmitriptan (2.5 mg/Day) (N=10) | Zolmitriptan (5 mg/Day) (N=11) | Zolmitriptan (10 mg/Day) (N=11)
Tachycardia (Cardiac disorders) | 5 | 4 | 3 | 5
Hypertension (Cardiac disorders) | 4 | 4 | 6 | 7
Deviated Midline Catheter (Surgical and medical procedures) | 2 | 0 | 0 | 0
ST Elevation More Peaked (Cardiac disorders) | 1 | 0 | 0 | 0
Tasting Saline (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Heartburn (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fever (Immune system disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Fluid Leak (from Midline) (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 (0) | 0 (0)
Pain at Midline Site (Skin and subcutaneous tissue disorders) | 0 (0) | 3 | 0 (0) | 1
Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 | 0 (0) | 0 (0)
Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 | 1
Skin Irritation from Adhesive (Skin and subcutaneous tissue disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Itching at Midline Site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1
Headache (Nervous system disorders) | 5 | 3 | 3 | 3
Sleepiness (Nervous system disorders) | 0 (0) | 1 | 0 (0) | 0 (0)
Sinus Headache (Nervous system disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 2 | 1 | 2 | 1
Vivid dreams (Nervous system disorders) | 1 | 0 (0) | 0 (0) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1
Diffuse body pain (Musculoskeletal and connective tissue disorders) | 1 | 0 (0) | 0 (0) | 1
foot pain (Musculoskeletal and connective tissue disorders) | 1 | 0 (0) | 0 (0) | 0 (0)
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT05019430/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT05019430/ICF_000.pdf